CLINICAL TRIAL: NCT03092791
Title: A Randomized, Observer-Blind, Controlled Phase 1/2 Trial to Evaluate the Safety, Tolerability and Immunogenicity of Different Doses of a Stand-alone Trivalent, Inactivated Poliomyelitis Vaccine From Sabin Strains in Healthy Infants, With a Safety and Tolerability Age-Step Down Lead-in in Healthy Adults Followed by Healthy Toddlers
Brief Title: IPV-102 Safety, Tolerability and Immunogenicity of TAK-195 in Healthy Infants, Toddlers and Adults
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Planned immunogenicity outcomes not reached
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPV-102; U1111-1191-6847 (Registry Identifier: World Health Organisation)
Record Dates: First submitted 2017-03-24; First posted 2017-03-28 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis
Keywords: Drug Therapy
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adult Lead-in Cohort: sIPV High Dose (Experimental): Sabin-based inactivated poliomyelitis vaccine (sIPV) containing 3, 100, and 100 D-Ag units (DU) of poliovirus types 1, 2, and 3, intramuscular injection on Day 1.
  Interventions: Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV)
- Adult Lead-in Cohort: Placebo (Placebo Comparator): Placebo, intramuscular injection on Day 1.
  Interventions: Biological: sIPV Placebo
- Toddler Lead-in Cohort: sIPV High Dose (Experimental): sIPV containing 3, 100, and 100 DU of poliovirus types 1, 2, and 3, intramuscular injection on Day 1.
  Interventions: Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV)
- Toddler Lead-in Cohort: Reference IPV (Active Comparator): Reference IPV, intramuscular injection on Day 1.
  Interventions: Biological: Reference IPV
- Infant Dose Ranging Cohort: sIPV Low Dose (Experimental): sIPV containing 0.75, 25, 25 DU of poliovirus types 1, 2, and 3, intramuscular injection on Days 1, 29, 57 and 365.
  Interventions: Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV)
- Infant Dose Ranging Cohort: sIPV Medium Dose (Experimental): sIPV containing 1.5, 50, 50 DU of poliovirus types 1, 2, and 3, intramuscular injection on Days 1, 29 57 and 365.
  Interventions: Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV)
- Infant Dose Ranging Cohort: sIPV High Dose (Experimental): sIPV containing 3, 100, 100 DU of poliovirus types 1, 2, and 3, intramuscular injection on Days 1, 29 57 and 365.
  Interventions: Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV)
- Infant Dose Ranging Cohort: Reference IPV (Active Comparator): Reference IPV, intramuscular injection on Days 1, 29 57 and 365.
  Interventions: Biological: Reference IPV

INTERVENTIONS:
Biological: Sabin-Based Inactivated Poliomyelitis Vaccine (sIPV) — sIPV intramuscular injection
  Arms: Adult Lead-in Cohort: sIPV High Dose; Infant Dose Ranging Cohort: sIPV High Dose; Infant Dose Ranging Cohort: sIPV Low Dose; Infant Dose Ranging Cohort: sIPV Medium Dose; Toddler Lead-in Cohort: sIPV High Dose
Biological: Reference IPV — Reference IPV intramuscular injection
  Arms: Infant Dose Ranging Cohort: Reference IPV; Toddler Lead-in Cohort: Reference IPV
Biological: sIPV Placebo — sIPV placebo-matching intramuscular injection
  Arms: Adult Lead-in Cohort: Placebo

SUMMARY:
The purpose of this study is to select the optimal antigen dosage of the three Sabin poliovirus strains (types 1, 2, and 3) entering the composition of the stand-alone trivalent Sabin-based inactivated poliomyelitis vaccine (sIPV) to take forward into advanced stage studies. The selection will be carried out comparing the three sIPV study arms based on the safety and tolerability profile after each dose of primary immunization and the immune response to poliovirus types 1, 2, and 3 for both Sabin and Salk strains, after the final dose of a three dose primary immunization series (Day 85).

DETAILED DESCRIPTION:
The vaccine being tested in this study is called sIPV. sIPV is used to prevent poliomyelitis. This study will look at the safety, tolerability of sIPV in healthy adults, toddlers and infants as well as safety and immunogenicity in toddlers and infants. .

The study will enroll approximately 340 participants including 40 adults, 60 toddlers and 240 infants. Adult participants will be randomly assigned to one of the two treatment groups-which will remain undisclosed to study doctor and participants during the study (unless there is an urgent medical need):

* sIPV High Dose
* Placebo (saline control - 0.9% sodium chloride)

Toddler participants will be randomly assigned to one of the following treatment groups:

* sIPV High Dose
* Reference IPV

Infant participants will be randomly assigned to one of following treatment groups:

* sIPV Low Dose
* sIPV Medium Dose
* sIPV High Dose
* Reference IPV Adults and toddlers will receive intramuscular injection on Day 1. Infants will receive intramuscular injection on Days 1, 29, 57 and 365.

This is a multicentre trial. The overall time to participate in this study for adult is 8 days, for toddlers is 183 days and infants is 547 days.

ELIGIBILITY:
Inclusion Criteria:

Adult Lead-in Cohort

1. Individuals who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
2. Completed primary immunization against poliomyelitis according to local recommendations.

Toddler Lead-in Cohort

1. Toddlers in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
2. Completed primary immunization against poliomyelitis, preferably with IPV, according to local recommendations.

Infant Dose Ranging Cohort 1. Infants are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.

3. Infants must have been born full term (37-42 weeks of gestation).

Exclusion Criteria:

Adult Lead-in Cohort

1. Has body mass index (BMI) greater than or equal to 35 kg/m^2 (= weight in kg [height in meters * height in meters].

Toddler Lead-in Cohort

1. Last polio vaccination (either inactivated or oral) received within 5 months prior to first trial visit.
2. Household member/sibling who had received or is/are scheduled to receive Oral Poliomyelitis Vaccine (OPV) in the previous 3 months until 5 weeks post participant's inclusion in the study.
3. Prior vaccination with booster dose of diphtheria, tetanus, pertussis (acellular or whole cell), polio (either inactivated or oral), or Haemophilus influenzae type b (Hib) vaccines.

Infant Dose Ranging Cohort

1. Infants with low birth weight according to local standards.
2. Prior vaccination with polio vaccines (either inactivated or oral).
3. Household member/sibling that had received or is/are scheduled to receive OPV in the previous 3 months until 5 weeks after the third dose of the primary immunization series.
4. Prior vaccination with any diphtheria, tetanus, pertussis (acellular or whole cell), Haemophilus influenzae type b (Hib) vaccine or polio vaccine (OPV or IPV). Note, bacillus Calmette Guérin (BCG) at birth and prior vaccination with Hepatitis B vaccine given at least 4 weeks prior to first trial visit are not exclusion criteria.

All Cohorts

1. Any significant chronic infection.
2. Any clinically significant active infection (as assessed by the investigator) or temperature ≥38.0°C (>100.4°F), within 3 days of intended trial vaccination.
3. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone for ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1.
   3. Administration of immunoglobulins and/or any blood or blood products within the 3 months preceding the administration of the trial vaccine or planned administration during the trial
   4. Receipt of immunostimulants within 60 days prior to Day 1.
   5. Genetic immunodeficiency.
4. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.

Ages: 6 Weeks to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 340 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director Clinical Science, Study Director — Takeda
Locations (4):
- Panama (4):
  - CEVAXIN - David, Chiriquí
  - CEVAXIN - 24 de Diciembre, Panama City
  - CEVAXIN - Chorrera, Panama City
  - CEVAXIN Plaza Carolina - Ciudad de Panama, Panama City

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at four investigative sites in Panama from 7 June 2017 to 18 October 2018.
Pre-assignment Details: Healthy participants were randomized to one of two (adult and toddler lead-ins) or four (infant dose ranging) arms in a 1:1 or a 1:1:1:1 ratio, to receive sIPV or reference sIPV. Two groups received placebo.
Groups:
- Infant Dose Ranging Cohort: sIPV Medium Dose: sIPV containing 1.5, 50, 50 DU of poliovirus types 1, 2, and 3, intramuscular injection on Days 1, 29, 57 and 365.
- Infant Dose Ranging Cohort: sIPV High Dose: sIPV containing 3, 100, 100 DU of poliovirus types 1, 2, and 3, intramuscular injection on Days 1, 29, 57 and 365.
- Infant Dose Ranging Cohort: Reference IPV: Reference IPV, intramuscular injection on Days 1, 29, 57 and 365.
Period: Overall Study
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Started | 20 | 20 | 30 | 30 | 60 | 60 | 60 | 60
Completed | 20 | 20 | 30 | 30 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 60 | 60 | 60 | 60
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 4 | 12 | 6 | 4
Not completed — Study Termination | 0 | 0 | 0 | 0 | 55 | 46 | 53 | 55
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV | Total
Number analyzed (Participants) | 20 | 20 | 30 | 30 | 60 | 60 | 60 | 60 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data for age in adults is reported.
  years
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 40
    (all) | 34.9 (8.56) | 35.1 (8.23) |  |  |  |  |  |  | 35.0 (8.29)
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: Data for age in toddlers is reported.
  months
    number analyzed (Participants) | 0 | 0 | 30 | 30 | 0 | 0 | 0 | 0 | 60
    (all) |  |  | 14.1 (0.98) | 14.0 (1.02) |  |  |  |  | 14.0 (0.99)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Population: Data for age in infants is reported.
  weeks
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 60 | 60 | 60 | 60 | 240
    (all) |  |  |  |  | 6.6 (0.67) | 6.5 (0.62) | 6.5 (0.68) | 6.5 (0.62) | 6.5 (0.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 13 | 12 | 31 | 33 | 29 | 22 | 169
  Male | 4 | 7 | 17 | 18 | 29 | 27 | 31 | 38 | 171
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 13 | 29 | 29 | 58 | 57 | 55 | 58 | 317
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 1 | 1 | 1 | 2 | 2 | 2 | 16
  White | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 6
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Panama | 20 | 20 | 30 | 30 | 60 | 60 | 60 | 60 | 340
Height [Mean (Full Range); unit: centimeter (cm)] | 160.00 [147.0 to 178.0] | 161.45 [149.0 to 189.0] | 77.13 [72.0 to 85.0] | 76.53 [70.0 to 80.0] | 55.71 [35.8 to 63.0] | 56.29 [52.0 to 72.0] | 55.21 [36.3 to 60.0] | 56.21 [51.0 to 75.0] | 87.31 [51.0 to 189.0]
Weight [Mean (Full Range); unit: kilogram (kg)] | 74.30 [56.5 to 100.0] | 68.74 [41.5 to 98.0] | 10.21 [8.4 to 12.5] | 10.32 [7.5 to 15.3] | 4.94 [3.7 to 6.6] | 4.94 [3.4 to 6.1] | 4.89 [3.6 to 6.3] | 4.98 [3.2 to 5.9] | 22.91 [3.2 to 100.0]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/[height (m)^2] Population: Data for BMI in adults is reported.
  kg/m^2
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 40
    (all) | 28.95 (3.253) | 26.25 (4.489) |  |  |  |  |  |  | 27.60 (4.103)
Baseline Seropositivity [Number; unit: percentage of participants seropositive] — Seropositivity defined as the percentage of participants with antibody titers ≥ 8. Population: Randomized set included all randomized participants. Number analyzed is the number of participants with data available for analysis at the given timepoint. Data are reported for 'Toddler Lead-in Cohort and Infant Dose Ranging Cohort'.
  percentage of participants seropositive
    Sabin Type 1: number analyzed (Participants) | 0 | 0 | 27 | 26 | 30 | 30 | 21 | 26 | 160
    Sabin Type 1 |  |  | 90.0 | 86.7 | 50.0 | 50.0 | 35.0 | 43.3 | 59.16
    Sabin Type 2: number analyzed (Participants) | 0 | 0 | 28 | 28 | 40 | 41 | 38 | 40 | 215
    Sabin Type 2 |  |  | 93.3 | 93.3 | 66.7 | 68.3 | 63.3 | 66.7 | 75.26
    Sabin Type 3: number analyzed (Participants) | 0 | 0 | 28 | 27 | 14 | 19 | 18 | 20 | 126
    Sabin Type 3 |  |  | 93.3 | 90.0 | 23.3 | 31.7 | 30.0 | 33.3 | 50.26
    Salk Type 1: number analyzed (Participants) | 0 | 0 | 29 | 29 | 20 | 22 | 18 | 20 | 138
    Salk Type 1 |  |  | 96.7 | 96.7 | 33.3 | 36.7 | 30.0 | 33.3 | 54.45
    Salk Type 2: number analyzed (Participants) | 0 | 0 | 29 | 27 | 24 | 26 | 25 | 24 | 155
    Salk Type 2 |  |  | 96.7 | 90.0 | 40.0 | 43.3 | 41.7 | 40.0 | 58.61
    Salk Type 3: number analyzed (Participants) | 0 | 0 | 28 | 27 | 13 | 9 | 14 | 13 | 104
    Salk Type 3 |  |  | 93.3 | 90.0 | 21.7 | 15.0 | 23.3 | 21.7 | 44.16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After First Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 1
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment, severe: prevents daily activity with or without treatment), erythema, induration and swelling (any: <25 mm, mild: >25 - ≤ 50 mm, moderate: > 50 - ≤ 100 mm, severe: > 100 mm). Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of the First Dose given on Day 1
Population: Safety Set in 'Infant Dose Ranging Cohort - sIPV arms' included all participants who received at least one dose of the trial vaccines. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Pain: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 56
  Pain: First Dose (Day 1), Any | 84.2 | 69.2 | 80.4
  Pain: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 56
  Pain: First Dose (Day 1), Mild | 26.3 | 30.8 | 41.1
  Pain: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 56
  Pain: First Dose (Day 1), Moderate | 31.6 | 17.3 | 25.0
  Pain: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 56
  Pain: First Dose (Day 1), Severe | 26.3 | 21.2 | 14.3
  Erythema: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 56
  Erythema: First Dose (Day 1), Any | 5.3 | 1.9 | 0
  Induration: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 51 | 56
  Induration: First Dose (Day 1), Any | 1.8 | 3.9 | 0
  Induration: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 51 | 56
  Induration: First Dose (Day 1), Moderate | 0 | 2.0 | 0
  Swelling: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 51 | 56
  Swelling: First Dose (Day 1), Any | 1.8 | 7.8 | 0
  Swelling: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 51 | 56
  Swelling: First Dose (Day 1), Moderate | 0 | 2.0 | 0

2. Primary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After Second Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 29
Description: as for outcome 1
Time Frame: Within 7 days of the Second Dose given on Day 29
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Pain: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Pain: Second Dose (Day 29), Any | 48.2 | 47.9 | 61.8
  Pain: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55
  Pain: Second Dose (Day 29), Mild | 30.4 | 25.0 | 36.4
  Pain: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55
  Pain: Second Dose (Day 29), Moderate | 14.3 | 16.7 | 18.2
  Pain: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55
  Pain: Second Dose (Day 29), Severe | 3.6 | 6.3 | 7.3
  Erythema: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Erythema: Second Dose (Day 29), Any | 1.8 | 2.1 | 0
  Induration: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Induration: Second Dose (Day 29), Any | 0 | 2.1 | 0
  Swelling: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Swelling: Second Dose (Day 29), Any | 0 | 4.2 | 0
  Swelling: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55
  Swelling: Second Dose (Day 29), Mild | 0 | 2.1 | 0

3. Primary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After Third Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 57
Description: as for outcome 1
Time Frame: Within 7 Days of the Third Dose given on Day 57
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Pain: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 45 | 53
  Pain: Third Dose (Day 57), Any | 46.4 | 44.4 | 49.1
  Pain: Third Dose (Day 57), Mild: number analyzed (Participants) | 56 | 45 | 53
  Pain: Third Dose (Day 57), Mild | 33.9 | 31.1 | 34.0
  Pain: Third Dose (Day 57), Moderate: number analyzed (Participants) | 56 | 45 | 53
  Pain: Third Dose (Day 57), Moderate | 8.9 | 8.9 | 11.3
  Pain: Third Dose (Day 57), Severe: number analyzed (Participants) | 56 | 45 | 53
  Pain: Third Dose (Day 57), Severe | 3.6 | 4.4 | 3.8
  Erythema: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 46 | 53
  Erythema: Third Dose (Day 57), Any | 0 | 2.2 | 1.9
  Swelling: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 46 | 53
  Swelling: Third Dose (Day 57), Any | 1.8 | 0 | 0

4. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Within 7-day Period (Including Day of Vaccination) After First Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 1
Description: Solicited systemic AEs were collected within 7 days after vaccination using a diary and included drowsiness, graded as 0-behavior as usual, 1-mild: drowsiness easily tolerated, 2-moderate: drowsiness that interferes with normal activity and 3-severe: prevents normal activity with or without treatment; irritability/fussiness, graded as 0-behavior as usual, mild: crying more than usual/no effect on normal activity, moderate: crying more than usual/interferes with normal activity and severe: crying that cannot be comforted/prevents normal; loss of appetite, graded as 0-apetite as usual, mild: eating less than usual/no effect on normal activity, moderate: eating less than usual/interferes with normal activity and severe: not eating at all. Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of the First Dose given on Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Drowsiness: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55
  Drowsiness: First Dose (Day 1), Any | 49.1 | 48.1 | 47.3
  Drowsiness: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55
  Drowsiness: First Dose (Day 1), Mild | 38.6 | 32.7 | 23.6
  Drowsiness: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55
  Drowsiness: First Dose (Day 1), Moderate | 8.8 | 13.5 | 21.8
  Drowsiness: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 55
  Drowsiness: First Dose (Day 1), Severe | 1.8 | 1.9 | 1.8
  Irritability: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55
  Irritability: First Dose (Day 1), Any | 56.1 | 57.7 | 58.2
  Irritability: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55
  Irritability: First Dose (Day 1), Mild | 28.1 | 28.8 | 29.1
  Irritability: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55
  Irritability: First Dose (Day 1), Moderate | 21.1 | 19.2 | 18.2
  Irritability: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 55
  Irritability: First Dose (Day 1), Severe | 7.0 | 9.6 | 10.9
  Loss of Appetite: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55
  Loss of Appetite: First Dose (Day 1), Any | 29.8 | 25.0 | 21.8
  Loss of Appetite: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55
  Loss of Appetite: First Dose (Day 1), Mild | 26.3 | 23.1 | 9.1
  Loss of Appetite: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55
  Loss of Appetite: First Dose (Day 1), Moderate | 3.5 | 1.9 | 12.7

5. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Within 7-day Period (Including Day of Vaccination) After Second Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 29
Description: as for outcome 4
Time Frame: Within 7 days of the Second Dose given on Day 29
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Drowsiness: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Drowsiness: Second Dose (Day 29), Any | 30.4 | 20.8 | 36.4
  Drowsiness: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55
  Drowsiness: Second Dose (Day 29), Mild | 19.6 | 18.8 | 25.5
  Drowsiness: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55
  Drowsiness: Second Dose (Day 29), Moderate | 10.7 | 2.1 | 10.9
  Irritability: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Irritability: Second Dose (Day 29), Any | 37.5 | 33.3 | 45.5
  Irritability: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55
  Irritability: Second Dose (Day 29), Mild | 19.6 | 25.0 | 30.9
  Irritability: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55
  Irritability: Second Dose (Day 29), Moderate | 10.7 | 6.3 | 9.1
  Irritability: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55
  Irritability: Second Dose (Day 29), Severe | 7.1 | 2.1 | 5.5
  Loss of Appetite: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55
  Loss of Appetite: Second Dose (Day 29), Any | 14.3 | 10.4 | 18.2
  Loss of Appetite: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55
  Loss of Appetite: Second Dose (Day 29), Mild | 12.5 | 8.3 | 16.4
  Loss of Appetite: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55
  Loss of Appetite: Second Dose (Day 29), Moderate | 1.8 | 2.1 | 0
  Loss of Appetite: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55
  Loss of Appetite: Second Dose (Day 29), Severe | 0 | 0 | 1.8

6. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Within 7-day Period (Including Day of Vaccination) After Third Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort by Severity on Day 57
Description: as for outcome 4
Time Frame: Within 7 Days of the Third Dose given on Day 57
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Drowsiness: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53
  Drowsiness: Third Dose (Day 57), Any | 38.2 | 21.7 | 32.1
  Drowsiness: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53
  Drowsiness: Third Dose (Day 57), Mild | 25.5 | 21.7 | 26.4
  Drowsiness: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53
  Drowsiness: Third Dose (Day 57), Moderate | 12.7 | 0 | 5.7
  Irritability: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53
  Irritability: Third Dose (Day 57), Any | 40.0 | 26.1 | 37.7
  Irritability: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53
  Irritability: Third Dose (Day 57), Mild | 27.3 | 21.7 | 28.3
  Irritability: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53
  Irritability: Third Dose (Day 57), Moderate | 5.5 | 2.2 | 7.5
  Irritability: Third Dose (Day 57), Severe: number analyzed (Participants) | 55 | 46 | 53
  Irritability: Third Dose (Day 57), Severe | 7.3 | 2.2 | 1.9
  Loss of Appetite: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53
  Loss of Appetite: Third Dose (Day 57), Any | 10.9 | 6.5 | 13.2
  Loss of Appetite: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53
  Loss of Appetite: Third Dose (Day 57), Mild | 9.1 | 6.5 | 13.2
  Loss of Appetite: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53
  Loss of Appetite: Third Dose (Day 57), Moderate | 1.8 | 0 | 0

7. Primary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After First Primary Immunization Dose of sIPV on Day 1
Description: A systemic adverse event (AE) of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 7 days after each Immunization. Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of the First Dose given on Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Fever: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55
  Fever: First Dose (Day 1), Any | 15.8 | 17.3 | 23.6
  Fever: First Dose (Day 1), 38.0°C - 38.4°C: number analyzed (Participants) | 57 | 52 | 55
  Fever: First Dose (Day 1), 38.0°C - 38.4°C | 8.8 | 9.6 | 14.5
  Fever: First Dose (Day 1), 38.5°C - 38.9°C: number analyzed (Participants) | 57 | 52 | 55
  Fever: First Dose (Day 1), 38.5°C - 38.9°C | 7.0 | 7.7 | 9.1

8. Primary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After Second Primary Immunization Dose of sIPV on Day 29
Description: A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 7 days after each Immunization. Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of the Second Dose given on Day 29
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Fever: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 47 | 54
  Fever: Second Dose (Day 29), Any | 7.1 | 6.4 | 14.8
  Fever: Second Dose (Day 29), 38.0°C - 38.4°C: number analyzed (Participants) | 56 | 47 | 54
  Fever: Second Dose (Day 29), 38.0°C - 38.4°C | 3.6 | 2.1 | 11.1
  Fever: Second Dose (Day 29), 38.5°C - 38.9°C: number analyzed (Participants) | 56 | 47 | 54
  Fever: Second Dose (Day 29), 38.5°C - 38.9°C | 3.6 | 2.1 | 3.7
  Fever: Second Dose (Day 29), 39.0°C - 39.4°C: number analyzed (Participants) | 56 | 47 | 54
  Fever: Second Dose (Day 29), 39.0°C - 39.4°C | 0 | 2.1 | 0

9. Primary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After Third Primary Immunization Dose of sIPV on Day 57
Description: as for outcome 8
Time Frame: Within 7 days of the Third Dose given on Day 57
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants
  Fever: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 52
  Fever: Third Dose (Day 57), Any | 9.1 | 8.7 | 15.4
  Fever: Third Dose (Day 57), 38.0°C - 38.4°C: number analyzed (Participants) | 55 | 46 | 52
  Fever: Third Dose (Day 57), 38.0°C - 38.4°C | 9.1 | 6.5 | 3.8
  Fever: Third Dose (Day 57), 38.5°C - 38.9°C: number analyzed (Participants) | 55 | 46 | 52
  Fever: Third Dose (Day 57), 38.5°C - 38.9°C | 0 | 0 | 7.7
  Fever: Third Dose (Day 57), 39.0°C - 39.4°C: number analyzed (Participants) | 55 | 46 | 52
  Fever: Third Dose (Day 57), 39.0°C - 39.4°C | 0 | 2.2 | 1.9
  Fever: Third Dose (Day 57), 39.5°C - 39.9°C: number analyzed (Participants) | 55 | 46 | 52
  Fever: Third Dose (Day 57), 39.5°C - 39.9°C | 0 | 0 | 1.9

10. Primary Outcome: Percentage of Participants Experiencing Non-serious Unsolicited AEs Within the 28-day Period (Including Day of Vaccination) After Each Primary Immunization Dose of sIPV in Infant Dose Ranging Cohort
Description: An AE is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. Non-serious unsolicited AEs indicates any and all AEs (other than serious adverse events [SAEs]) that occurred other than those that are solicited.
Time Frame: Within 28 days of primary vaccinations given on Days 1, 29 and 57 (Up to Day 85)
Population: Safety Set in 'Infant Dose Ranging Cohort - sIPV arms' included all participants who received at least one dose of the trial vaccines.
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants | 28.8 | 28.3 | 31.7

11. Primary Outcome: Percentage of Participants Experiencing SAEs Throughout the Entire Trial Duration in the sIPV Study Arms in Infant Dose Ranging Cohort
Description: An SAE is defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Day 1 up to Day 547
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose
Number analyzed (Participants) | 59 | 60 | 60
percentage of participants | 13.6 | 8.3 | 8.3

12. Primary Outcome: Percentage of Participants With Seroconversion
Description: Seroconversion is defined as i) initially seronegative infants (titer <8 at Day 1) having a titer ≥8 at Day 85, or ii) initially seropositive infants (titer ≥8 at Day 1) with a 4-fold rise in antibody titers over the expected level of maternal antibodies at Day 85, calculated using a decline from the Day 1 titer with a half-life of 28 days.
Time Frame: Day 85
Population: Per-protocol set (PPS) in 'Infant Dose Ranging Cohort' included all participants in full analysis set (FAS) who had no major protocol violations. FAS included all participants who were randomized and received at least one dose of trial vaccines. Number analyzed is number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 56 | 47 | 54 | 55
percentage of participants
  Sabin Type 1: Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Sabin Type 1: Day 85 | 63.0 [48.7 to 75.7] | 77.8 [62.9 to 88.8] | 86.0 [73.3 to 94.2] | 92.5 [81.8 to 97.9]
  Sabin Type 2: Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Sabin Type 2: Day 85 | 68.5 [54.4 to 80.5] | 77.8 [62.9 to 88.8] | 90.0 [78.2 to 96.7] | 94.3 [84.3 to 98.8]
  Sabin Type 3, Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Sabin Type 3, Day 85 | 96.3 [87.3 to 99.5] | 100 [92.1 to 100] | 96.0 [86.3 to 99.5] | 96.2 [87.0 to 99.5]
  Salk Type 1: Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Salk Type 1: Day 85 | 37.0 [24.3 to 51.3] | 53.3 [37.9 to 68.3] | 68.0 [53.3 to 80.5] | 96.2 [87.0 to 99.5]
  Salk Type 2: Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Salk Type 2: Day 85 | 35.2 [22.7 to 49.4] | 55.6 [40.0 to 70.4] | 70.0 [55.4 to 82.1] | 96.2 [87.0 to 99.5]
  Salk Type 3: Day 85: number analyzed (Participants) | 54 | 45 | 50 | 53
  Salk Type 3: Day 85 | 90.7 [79.7 to 96.9] | 93.3 [81.7 to 98.6] | 94.0 [83.5 to 98.7] | 94.3 [84.3 to 98.8]

13. Secondary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After Each Primary Immunization Dose of sIPV or IPV by Severity in Infant Dose Ranging Cohort
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (0-none, 1-mild: Minor reaction to touch, 2-moderate: Cries/protests on touch, 3-severe: Cries when limb is moved/spontaneously painful), erythema, induration and swelling (0: <10 mm, 1-Mild: >10 - ≤ 20 mm, 2-Moderate: > 20 - ≤ 40 mm, 3-Severe: > 40 mm). Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of primary vaccinations (First Dose given on Day 1, Second Dose given on Day 29, Third Dose given on Day 57)
Population: Safety Set in 'Infant Dose Ranging Cohort' included all participants who received at least one dose of the trial vaccines. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 59 | 60 | 60 | 60
percentage of participants
  Pain: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 56 | 57
  Pain: First Dose (Day 1), Any | 84.2 | 69.2 | 80.4 | 86.0
  Pain: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 56 | 57
  Pain: First Dose (Day 1), Mild | 26.3 | 30.8 | 41.1 | 22.8
  Pain: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 56 | 57
  Pain: First Dose (Day 1), Moderate | 31.6 | 17.3 | 25.0 | 40.4
  Pain: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 56 | 57
  Pain: First Dose (Day 1), Severe | 26.3 | 21.2 | 14.3 | 22.8
  Erythema: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 56 | 57
  Erythema: First Dose (Day 1), Any | 5.3 | 1.9 | 0 | 1.8
  Induration: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 51 | 56 | 57
  Induration: First Dose (Day 1), Any | 1.8 | 3.9 | 0 | 1.8
  Induration: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 51 | 56 | 57
  Induration: First Dose (Day 1), Moderate | 0 | 2.0 | 0 | 0
  Swelling: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 51 | 56 | 57
  Swelling: First Dose (Day 1), Any | 1.8 | 7.8 | 0 | 1.8
  Swelling: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 51 | 56 | 57
  Swelling: First Dose (Day 1), Moderate | 0 | 2.0 | 0 | 0
  Pain: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Pain: Second Dose (Day 29), Any | 48.2 | 47.9 | 61.8 | 59.6
  Pain: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55 | 57
  Pain: Second Dose (Day 29), Mild | 30.4 | 25.0 | 36.4 | 45.6
  Pain: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55 | 57
  Pain: Second Dose (Day 29), Moderate | 14.3 | 16.7 | 18.2 | 8.8
  Pain: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55 | 57
  Pain: Second Dose (Day 29), Severe | 3.6 | 6.3 | 7.3 | 5.3
  Erythema: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Erythema: Second Dose (Day 29), Any | 1.8 | 2.1 | 0 | 0
  Induration: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Induration: Second Dose (Day 29), Any | 0 | 2.1 | 0 | 0
  Swelling: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Swelling: Second Dose (Day 29), Any | 0 | 4.2 | 0 | 0
  Swelling: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55 | 57
  Swelling: Second Dose (Day 29), Mild | 0 | 2.1 | 0 | 0
  Pain: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 45 | 53 | 56
  Pain: Third Dose (Day 57), Any | 46.4 | 44.4 | 49.1 | 60.7
  Pain: Third Dose (Day 57), Mild: number analyzed (Participants) | 56 | 45 | 53 | 56
  Pain: Third Dose (Day 57), Mild | 33.9 | 31.1 | 34.0 | 48.2
  Pain: Third Dose (Day 57), Moderate: number analyzed (Participants) | 56 | 45 | 53 | 56
  Pain: Third Dose (Day 57), Moderate | 8.9 | 8.9 | 11.3 | 8.9
  Pain: Third Dose (Day 57), Severe: number analyzed (Participants) | 56 | 45 | 53 | 56
  Pain: Third Dose (Day 57), Severe | 3.6 | 4.4 | 3.8 | 3.6
  Erythema: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 46 | 53 | 56
  Erythema: Third Dose (Day 57), Any | 0 | 2.2 | 1.9 | 1.8
  Induration: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 46 | 53 | 56
  Induration: Third Dose (Day 57), Any | 0 | 0 | 0 | 1.8
  Swelling: Third Dose (Day 57), Any: number analyzed (Participants) | 56 | 46 | 53 | 56
  Swelling: Third Dose (Day 57), Any | 1.8 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Within 7-day Period (Including Day of Vaccination) After Each Primary Immunization Dose of sIPV or IPV by Severity in Infant Dose Ranging Cohort
Description: as for outcome 4
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 59 | 60 | 60 | 60
percentage of participants
  Drowsiness: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55 | 56
  Drowsiness: First Dose (Day 1), Any | 49.1 | 48.1 | 47.3 | 44.6
  Drowsiness: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55 | 56
  Drowsiness: First Dose (Day 1), Mild | 38.6 | 32.7 | 23.6 | 26.8
  Drowsiness: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55 | 56
  Drowsiness: First Dose (Day 1), Moderate | 8.8 | 13.5 | 21.8 | 16.1
  Drowsiness: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 55 | 56
  Drowsiness: First Dose (Day 1), Severe | 1.8 | 1.9 | 1.8 | 1.8
  Irritability: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55 | 57
  Irritability: First Dose (Day 1), Any | 56.1 | 57.7 | 58.2 | 61.4
  Irritability: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55 | 57
  Irritability: First Dose (Day 1), Mild | 28.1 | 28.8 | 29.1 | 28.1
  Irritability: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55 | 57
  Irritability: First Dose (Day 1), Moderate | 21.1 | 19.2 | 18.2 | 22.8
  Irritability: First Dose (Day 1), Severe: number analyzed (Participants) | 57 | 52 | 55 | 57
  Irritability: First Dose (Day 1), Severe | 7.0 | 9.6 | 10.9 | 10.5
  Loss of Appetite: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55 | 57
  Loss of Appetite: First Dose (Day 1), Any | 29.8 | 25.0 | 21.8 | 19.3
  Loss of Appetite: First Dose (Day 1), Mild: number analyzed (Participants) | 57 | 52 | 55 | 57
  Loss of Appetite: First Dose (Day 1), Mild | 26.3 | 23.1 | 9.1 | 8.8
  Loss of Appetite: First Dose (Day 1), Moderate: number analyzed (Participants) | 57 | 52 | 55 | 57
  Loss of Appetite: First Dose (Day 1), Moderate | 3.5 | 1.9 | 12.7 | 10.5
  Drowsiness: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Drowsiness: Second Dose (Day 29), Any | 30.4 | 20.8 | 36.4 | 29.8
  Drowsiness: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55 | 57
  Drowsiness: Second Dose (Day 29), Mild | 19.6 | 18.8 | 25.5 | 22.8
  Drowsiness: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55 | 57
  Drowsiness: Second Dose (Day 29), Moderate | 10.7 | 2.1 | 10.9 | 7.0
  Irritability: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Irritability: Second Dose (Day 29), Any | 37.5 | 33.3 | 45.5 | 38.6
  Irritability: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55 | 57
  Irritability: Second Dose (Day 29), Mild | 19.6 | 25.0 | 30.9 | 26.3
  Irritability: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55 | 57
  Irritability: Second Dose (Day 29), Moderate | 10.7 | 6.3 | 9.1 | 8.8
  Irritability: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55 | 57
  Irritability: Second Dose (Day 29), Severe | 7.1 | 2.1 | 5.5 | 3.5
  Loss of Appetite: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 48 | 55 | 57
  Loss of Appetite: Second Dose (Day 29), Any | 14.3 | 10.4 | 18.2 | 8.8
  Loss of Appetite: Second Dose (Day 29), Mild: number analyzed (Participants) | 56 | 48 | 55 | 57
  Loss of Appetite: Second Dose (Day 29), Mild | 12.5 | 8.3 | 16.4 | 8.8
  Loss of Appetite: Second Dose (Day 29), Moderate: number analyzed (Participants) | 56 | 48 | 55 | 57
  Loss of Appetite: Second Dose (Day 29), Moderate | 1.8 | 2.1 | 0 | 0
  Loss of Appetite: Second Dose (Day 29), Severe: number analyzed (Participants) | 56 | 48 | 55 | 57
  Loss of Appetite: Second Dose (Day 29), Severe | 0 | 0 | 1.8 | 0
  Drowsiness: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53 | 56
  Drowsiness: Third Dose (Day 57), Any | 38.2 | 21.7 | 32.1 | 25.0
  Drowsiness: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53 | 56
  Drowsiness: Third Dose (Day 57), Mild | 25.5 | 21.7 | 26.4 | 16.1
  Drowsiness: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53 | 56
  Drowsiness: Third Dose (Day 57), Moderate | 12.7 | 0 | 5.7 | 8.9
  Irritability: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53 | 56
  Irritability: Third Dose (Day 57), Any | 40.0 | 26.1 | 37.7 | 33.9
  Irritability: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53 | 56
  Irritability: Third Dose (Day 57), Mild | 27.3 | 21.7 | 28.3 | 26.8
  Irritability: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53 | 56
  Irritability: Third Dose (Day 57), Moderate | 5.5 | 2.2 | 7.5 | 7.1
  Irritability: Third Dose (Day 57), Severe: number analyzed (Participants) | 55 | 46 | 53 | 56
  Irritability: Third Dose (Day 57), Severe | 7.3 | 2.2 | 1.9 | 0
  Loss of Appetite: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 53 | 56
  Loss of Appetite: Third Dose (Day 57), Any | 10.9 | 6.5 | 13.2 | 8.9
  Loss of Appetite: Third Dose (Day 57), Mild: number analyzed (Participants) | 55 | 46 | 53 | 56
  Loss of Appetite: Third Dose (Day 57), Mild | 9.1 | 6.5 | 13.2 | 3.6
  Loss of Appetite: Third Dose (Day 57), Moderate: number analyzed (Participants) | 55 | 46 | 53 | 56
  Loss of Appetite: Third Dose (Day 57), Moderate | 1.8 | 0 | 0 | 3.6
  Loss of Appetite: Third Dose (Day 57), Severe: number analyzed (Participants) | 55 | 46 | 53 | 56
  Loss of Appetite: Third Dose (Day 57), Severe | 0 | 0 | 0 | 1.8

15. Secondary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After Each Primary Immunization Dose of sIPV or IPV in Infant Dose Ranging Cohort
Description: as for outcome 8
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 59 | 60 | 60 | 60
percentage of participants
  Fever: First Dose (Day 1), Any: number analyzed (Participants) | 57 | 52 | 55 | 57
  Fever: First Dose (Day 1), Any | 15.8 | 17.3 | 23.6 | 33.3
  Fever: First Dose (Day 1), 38.0°C - 38.4°C: number analyzed (Participants) | 57 | 52 | 55 | 57
  Fever: First Dose (Day 1), 38.0°C - 38.4°C | 8.8 | 9.6 | 14.5 | 15.8
  Fever: First Dose (Day 1), 38.5°C - 38.9°C: number analyzed (Participants) | 57 | 52 | 55 | 57
  Fever: First Dose (Day 1), 38.5°C - 38.9°C | 7.0 | 7.7 | 9.1 | 15.8
  Fever: First Dose (Day 1), >= 40.0°C: number analyzed (Participants) | 57 | 52 | 55 | 57
  Fever: First Dose (Day 1), >= 40.0°C | 0 | 0 | 0 | 1.8
  Fever: Second Dose (Day 29), Any: number analyzed (Participants) | 56 | 47 | 54 | 57
  Fever: Second Dose (Day 29), Any | 7.1 | 6.4 | 14.8 | 10.5
  Fever: Second Dose (Day 29), 38.0°C - 38.4°C: number analyzed (Participants) | 56 | 47 | 54 | 57
  Fever: Second Dose (Day 29), 38.0°C - 38.4°C | 3.6 | 2.1 | 11.1 | 7.0
  Fever: Second Dose (Day 29), 38.5°C - 38.9°C: number analyzed (Participants) | 56 | 47 | 54 | 57
  Fever: Second Dose (Day 29), 38.5°C - 38.9°C | 3.6 | 2.1 | 3.7 | 3.5
  Fever: Second Dose (Day 29), 39.0°C - 39.4°C: number analyzed (Participants) | 56 | 47 | 54 | 57
  Fever: Second Dose (Day 29), 39.0°C - 39.4°C | 0 | 2.1 | 0 | 0
  Fever: Third Dose (Day 57), Any: number analyzed (Participants) | 55 | 46 | 52 | 56
  Fever: Third Dose (Day 57), Any | 9.1 | 8.7 | 15.4 | 12.5
  Fever: Third Dose (Day 57), 38.0°C - 38.4°C: number analyzed (Participants) | 55 | 46 | 52 | 56
  Fever: Third Dose (Day 57), 38.0°C - 38.4°C | 9.1 | 6.5 | 3.8 | 7.1
  Fever: Third Dose (Day 57), 38.5°C - 38.9°C: number analyzed (Participants) | 55 | 46 | 52 | 56
  Fever: Third Dose (Day 57), 38.5°C - 38.9°C | 0 | 0 | 7.7 | 5.4
  Fever: Third Dose (Day 57), 39.0°C - 39.4°C: number analyzed (Participants) | 55 | 46 | 52 | 56
  Fever: Third Dose (Day 57), 39.0°C - 39.4°C | 0 | 2.2 | 1.9 | 0
  Fever: Third Dose (Day 57), 39.5°C - 39.9°C: number analyzed (Participants) | 55 | 46 | 52 | 56
  Fever: Third Dose (Day 57), 39.5°C - 39.9°C | 0 | 0 | 1.9 | 0

16. Secondary Outcome: Percentage of Participants Experiencing Non-serious Unsolicited AEs Within the 28-day Period (Including Day of Vaccination) After Each Primary Immunization Dose of sIPV or IPV in Infant Dose Ranging Cohort
Description: as for outcome 10
Time Frame: Within 28 Days of primary vaccinations (Up to 85 days)
Population: Safety Set in 'Infant Dose Ranging Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 59 | 60 | 60 | 60
percentage of participants | 28.8 | 28.3 | 31.7 | 33.3

17. Secondary Outcome: Percentage of Participants Experiencing SAEs Throughout the Entire Trial Duration in the sIPV or IPV Study Arms in Infant Dose Ranging Cohort
Description: as for outcome 11
Time Frame: Day 1 up to Day 547
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 59 | 60 | 60 | 60
percentage of participants | 13.6 | 8.3 | 8.3 | 13.3

18. Secondary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After Booster Vaccination in Infant Dose Ranging Cohort
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (0-none, 1-mild: Minor reaction to touch, 2-moderate: Cries/protests on touch, 3-severe: Cries when limb is moved/spontaneously painful), erythema, induration and swelling (0: <10 mm, 1-Mild: >10 - ≤ 20 mm, 2-Moderate: > 20 - ≤ 40 mm, 3-Severe: > 40 mm).
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Solicited Systemic AEs Within 7-day Period (Including Day of Vaccination) After Booster Vaccination in Infant Dose Ranging Cohort
Description: Percentage of participants with solicited systemic adverse events on a symptom by symptom basis, in each severity category will be reported. Solicited systemic adverse events include drowsiness, irritability/fussiness, loss of appetite, and fever. Fever is defined as greater than or equal to 38°C (100.4°F) regardless of method used.
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After Booster Vaccination in Infant Dose Ranging Cohort
Description: Fever is defined as greater than or equal to 38°C (100.4°F) regardless of method used.
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Percentage of Participants Experiencing Non-serious Unsolicited AEs Within the 28-day Period (Including Day of Vaccination) After Booster Vaccination in Infant Dose Ranging Cohort
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Non-serious unsolicited AEs indicates any and all AEs (other than SAEs) that occurred other than those that are solicited.
Time Frame: Within 28 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After Booster Vaccination in Toddler Lead-in Cohort
Description: Percentage of participants with solicited local reactions on a symptom by symptom basis, in each severity category will be reported. Solicited local reactions include pain, erythema, induration and swelling.
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percentage of Participants With Solicited Systemic AEs Within 7-day Period (Including Day of Vaccination) After Booster Vaccination in Toddler Lead-in Cohort
Description: Percentage of participants with solicited systemic adverse events on a symptom by symptom basis, in each severity category will be reported. Solicited systemic adverse events include headache, asthenia, malaise, arthralgia, myalgia.
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Percentage of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After Booster Vaccination in Toddler Lead-in Cohort
Description: Fever is defined as greater than or equal to 38°C (100.4°F) regardless of method used.
Time Frame: Within 7 days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Percentage of Participants Experiencing Non-serious Unsolicited AEs Within the 28-day Period (Including Day of Vaccination) After Booster Vaccination in Toddler Lead-in Cohort
Description: as for outcome 10
Time Frame: Within 28 Days of booster vaccination given on Day 365
Population: Study was terminated early, therefore data were not collected.
Arm/Group | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Percentage of Participants Experiencing SAEs Throughout the Entire Trial Duration in Toddler Lead-in Cohort
Description: as for outcome 11
Time Frame: Day 1 up to Day 183
Population: Safety Set in 'Toddlers Lead-in Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Number; unit: percentage of participants
Arm/Group | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV
Number analyzed (Participants) | 30 | 30
percentage of participants | 0 | 0

27. Secondary Outcome: Number of Participants With Solicited Local Reactions Within 7-day Period (Including Day of Vaccination) After a Single Dose of sIPV or Placebo in Adult Lead-in Cohort
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment, severe: prevents daily activity with or without treatment), erythema, induration and swelling (any: <25 mm, mild: >25 - ≤ 50 mm, moderate: > 50 - ≤ 100 mm, severe: > 100 mm).
Time Frame: Within 7 days of sIPV or placebo vaccination
Population: Safety Set in 'Adult Lead-in Cohort' included all participants who received at least one dose of the trial vaccines. Only categories for which there was at least 1 participant are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Pain: First Dose (Day 1), Any | 9 | 4
  Pain: First Dose (Day 1), Mild | 7 | 4
  Pain: First Dose (Day 1), Moderate | 2 | 0
  Erythema: First Dose (Day 1), Any | 1 | 0
  Induration: First Dose (Day 1), Any | 0 | 1
  Induration: First Dose (Day 1), Mild | 0 | 1
  Swelling: First Dose (Day 1), Any | 0 | 1
  Swelling: First Dose (Day 1), Mild | 0 | 1

28. Secondary Outcome: Number of Participants With Solicited Systemic AEs Within 7-day Period (Including Day of Vaccination) After a Single Dose of sIPV or Placebo in Adult Lead-in Cohort
Description: Solicited systemic AEs were collected by participants within 7 days after vaccination and included headache, asthenia, malaise, arthralgia and myalgia and fever. Severity scales for headache were none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents normal activity with or without treatment. Severity scales for others were none, mild: no interference with daily activity, moderate: interference with daily activity and severe: prevents daily activity. Data is only reported for those categories with at least 1 participant.
Time Frame: Within 7 days of sIPV or placebo vaccination
Population: Safety Set in 'Adult Lead-in Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Headache: First Dose (Day 1), Any | 3 | 3
  Headache: First Dose (Day 1), Mild | 1 | 3
  Headache: First Dose (Day 1), Moderate | 1 | 0
  Headache: First Dose (Day 1), Severe | 1 | 0
  Malaise: First Dose (Day 1), Any | 1 | 1
  Malaise: First Dose (Day 1), Mild | 0 | 1
  Malaise: First Dose (Day 1), Moderate | 1 | 0
  Arthralgia: First Dose (Day 1), Any | 4 | 3
  Arthralgia: First Dose (Day 1), Mild | 2 | 1
  Myalgia: First Dose (Day 1), Any | 4 | 3
  Myalgia: First Dose (Day 1), Mild | 2 | 2
  Myalgia: First Dose (Day 1), Moderate | 2 | 1

29. Secondary Outcome: Number of Participants With a Body Temperature ≥ 38°C (Defined as Fever) During the 7-day Period (Including Day of Vaccination) After a Single Dose of sIPV or Placebo in Adult Lead-in Cohort
Description: as for outcome 8
Time Frame: Within 7 days of sIPV or placebo vaccination dose given on Day 1
Population: Safety Set in 'Adult Lead-in Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Fever: First Dose (Day 1), Any | 0 | 1
  Fever: First Dose (Day 1), 38.5°C - 38.9°C | 0 | 1

30. Secondary Outcome: Number of Participants Experiencing Non-serious Unsolicited AEs Within the 7-day Period (Including Day of Vaccination) After a Single Dose of sIPV or Placebo in Adult Lead-in Cohort
Description: as for outcome 10
Time Frame: Within 7 days of sIPV or placebo vaccination
Population: Safety Set in 'Adult Lead-in Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

31. Secondary Outcome: Number of Participants Experiencing SAEs Throughout the Entire Trial Duration in Adult Lead-in Cohort
Description: as for outcome 11
Time Frame: Day 1 up to Day 8
Population: Safety Set in 'Adult Lead-in Cohort' included all participants who received at least one dose of the trial vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

32. Secondary Outcome: Seropositivity/Seroprotection Rate (SPR) on Days 85, 365 and 393 in Infant Dose Ranging Cohort
Description: SPR is defined as the percentage of participants with antibodies titers of poliovirus types 1, 2, and 3 for both Sabin and Salk strain ≥8.
Time Frame: Days 85, 365 and 393
Population: Per-protocol set (PPS) included all participants in the full analysis set (FAS) who had no major protocol violations. The FAS included all participants who were randomized and received at least one dose of the trial vaccines. Study was early terminated, thus data for Days 365 and 393 are not reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 56 | 47 | 54 | 55
percentage of participants
  Sabin Type 1: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 1: Day 85 | 72.2 [58.4 to 83.5] | 89.1 [76.4 to 96.4] | 88.0 [75.7 to 95.5] | 96.2 [87.0 to 99.5]
  Sabin Type 2: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 2: Day 85 | 83.3 [70.7 to 92.1] | 95.7 [85.2 to 99.5] | 100 [92.9 to 100] | 98.1 [89.9 to 100]
  Sabin Type 3: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 3: Day 85 | 98.1 [90.1 to 100] | 100 [92.3 to 100] | 98.0 [89.4 to 99.9] | 100 [93.3 to 100]
  Salk Type 1: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Salk Type 1: Day 85 | 42.6 [29.2 to 56.8] | 56.5 [41.1 to 71.1] | 72.0 [57.5 to 83.8] | 96.2 [87.0 to 99.5]
  Salk Type 2: Day 85: number analyzed (Participants) | 55 | 46 | 54 | 52
  Salk Type 2: Day 85 | 38.9 [25.9 to 53.1] | 65.2 [49.8 to 78.6] | 74.0 [59.7 to 85.4] | 100 [93.3 to 100]
  Salk Type 3: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Salk Type 3: Day 85 | 92.6 [82.1 to 97.9] | 93.5 [82.1 to 98.6] | 96.0 [86.3 to 99.5] | 98.1 [89.9 to 100]

33. Secondary Outcome: Geometric Mean Titers (GMT) on Days 85, 365 and 393 in Infant Dose Ranging Cohort
Description: GMT titers for poliovirus types 1, 2, and 3 for both Sabin and Salk strains will be reported.
Time Frame: Days 85, 365 and 393
Population: PPS in 'Infant Dose Ranging Cohort': participants in FAS who had no major protocol violations. FAS: participants who were randomized and received at least one dose of trial vaccines. Number analyzed is number of participants with data available for analysis at given timepoint. Study was early terminated, data for Days 365 and 393 are not reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 56 | 47 | 54 | 55
titer
  Sabin Type 1: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 1: Day 85 | 47.2 [28.2 to 78.8] | 105.6 [61.8 to 180.4] | 222.7 [130.6 to 379.7] | 155.0 [104.4 to 230.3]
  Sabin Type 2: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 2: Day 85 | 53.2 [34.4 to 82.3] | 119.7 [74.2 to 192.9] | 205.1 [138.9 to 303.0] | 268.1 [188.4 to 381.5]
  Sabin Type 3: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Sabin Type 3: Day 85 | 400.0 [267.3 to 598.4] | 748.2 [540.5 to 1035.7] | 844.6 [598.2 to 1192.5] | 533.8 [391.8 to 727.1]
  Salk Type 1: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Salk Type 1: Day 85 | 11.7 [8.6 to 15.7] | 18.2 [11.5 to 28.9] | 27.5 [17.8 to 42.6] | 719.4 [520.9 to 993.7]
  Salk Type 2: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Salk Type 2: Day 85 | 14.3 [9.7 to 21.2] | 22.4 [14.8 to 33.9] | 26.2 [18.2 to 37.6] | 400.1 [296.7 to 539.7]
  Salk Type 3: Day 85: number analyzed (Participants) | 54 | 46 | 50 | 53
  Salk Type 3: Day 85 | 139.7 [83.7 to 233.2] | 257.9 [160.0 to 415.6] | 361.2 [230.4 to 566.2] | 456.2 [317.3 to 656.0]

34. Secondary Outcome: Vaccine Response Rate (VRR) on Day 393 in Infant Dose Ranging Cohort
Description: VRR is defined as percentage of participants i) seronegative prior to booster vaccination (titer <8) having a titer ≥8, or ii) seropositive prior to booster vaccination (titer ≥8) having a 4-fold rise in antibody titers.
Time Frame: Day 393
Population: As the study was early terminated the data was not collected at Day 393 for Vaccine Response Rate.
Arm/Group | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 8 for Adults, Day 183 for Toddlers and Day 597 for Infants
Description: At each visit the investigator had to document any occurrence of non-serious adverse events and SAEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Adult Lead-in Cohort: sIPV High Dose | Adult Lead-in Cohort: Placebo | Toddler Lead-in Cohort: sIPV High Dose | Toddler Lead-in Cohort: Reference IPV | Infant Dose Ranging Cohort: sIPV Low Dose | Infant Dose Ranging Cohort: sIPV Medium Dose | Infant Dose Ranging Cohort: sIPV High Dose | Infant Dose Ranging Cohort: Reference IPV
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/30 | 0/30 | 0/59 | 1/60 | 0/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/30 | 0/30 | 8/59 | 5/60 | 5/60 | 8/60
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 8/30 | 13/30 | 17/59 | 17/60 | 19/60 | 20/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Lead-in Cohort: sIPV High Dose (N=20) | Adult Lead-in Cohort: Placebo (N=20) | Toddler Lead-in Cohort: sIPV High Dose (N=30) | Toddler Lead-in Cohort: Reference IPV (N=30) | Infant Dose Ranging Cohort: sIPV Low Dose (N=59) | Infant Dose Ranging Cohort: sIPV Medium Dose (N=60) | Infant Dose Ranging Cohort: sIPV High Dose (N=60) | Infant Dose Ranging Cohort: Reference IPV (N=60)
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One death occurred during treatment and was not related.
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One death occurred during treatment and was not related
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Lead-in Cohort: sIPV High Dose (N=20) | Adult Lead-in Cohort: Placebo (N=20) | Toddler Lead-in Cohort: sIPV High Dose (N=30) | Toddler Lead-in Cohort: Reference IPV (N=30) | Infant Dose Ranging Cohort: sIPV Low Dose (N=59) | Infant Dose Ranging Cohort: sIPV Medium Dose (N=60) | Infant Dose Ranging Cohort: sIPV High Dose (N=60) | Infant Dose Ranging Cohort: Reference IPV (N=60)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 5 | 8 | 9 | 9 | 13 | 13
Influenza (Infections and infestations) | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 7 | 7 | 4 | 5
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT03092791/SAP_000.pdf
  • Study Protocol (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03092791/Prot_001.pdf